CLINICAL TRIAL: NCT04337528
Title: Biomechanical Effects of Osteopathic Thrust and Muscle-energy Manipulations in Sacroiliac Joint Dysfunction of Athletes or Runners
Brief Title: Osteopathic Thrust and Muscle-energy Manipulations on Sacroiliac Joint Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Linda H. Chung, Contracted Professor (Contratado Doctor), Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE031911
Record Dates: First submitted 2020-02-18; First posted 2020-04-07 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Sacroiliac Disorder
Keywords: osteopathy; baropodometry

STUDY DESIGN:
Intervention Model Description: Group 1: Thrust technique Group 2: Muscle-energy technique Group 3: Placebo
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the assessor of pre-post-biomechanical measurements will be blinded to which manipulation the participant has been assigned to. The manipulation intervention will be performed by a separate physical therapist who is not involved with the biomechanical measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thrust Group (Experimental): Participant will receive the thrust technique manipulation of the affected sacroiliac joint.
  Interventions: Other: Osteopathic manipulation type muscle-energy; Other: Placebo technique
- Muscle-energy group (Active Comparator): Participant will receive the muscle-energy technique manipulation of the affected sacroiliac joint.
  Interventions: Other: Osteopathic manipulation type thrust; Other: Placebo technique
- Placebo Group (Placebo Comparator): Participant will receive a placebo manipulation of the affected sacroiliac joint.
  Interventions: Other: Osteopathic manipulation type thrust; Other: Osteopathic manipulation type muscle-energy

INTERVENTIONS:
Other: Osteopathic manipulation type thrust — The osteopathic manipulation type thrust is applied to solve the sacroiliac joint dysfunction. This technique applies a high velocity and intensity push in a specified direction to correct the dysfunction produced by a not correct position or movement of one joint.
  Arms: Muscle-energy group; Placebo Group
Other: Osteopathic manipulation type muscle-energy — The muscle-energy manipulation is applied to solve the sacroiliac joint dysfunction. This technique applies a movement with an intermittent resistance in a specified direction to correct the position or movement of one joint. The therapist applies the movement in the correct direction since he feels a limitation of movement. When he feels the limitation he requests to the participant pushing in the contrary direction without movement. After five or seven seconds the participant finishes the contraction and the therapist continues the correct movement since he feels once again the limitation, and he request to the participant contraction another five or seven seconds. The therapist request to the participant only three times, when he finish the three contraction and the therapy applies the last movement to correct direction the intervention finishes.
  Arms: Placebo Group; Thrust Group
Other: Placebo technique — The therapist simulates a false technique. The therapist applies movement in the sacroiliac joint without dysfunction, he applies movement since ninety degrees of pelvic flexion, and he wait sixty seconds. Whit this placebo technique the sacroiliac joint with the dysfunction is not altered.
  Arms: Muscle-energy group; Thrust Group

SUMMARY:
This study assesses the effect of manipulative techniques of thrust and muscle-energy over the sacroiliac joint on plantar foot support, weight distribution in the lower limbs and balance in amateur runners with sacroiliac dysfunction. participants will be randomly assigned to one of 3 manipulations (i.e., intervention): thrust, muscle-energy or placebo.

DETAILED DESCRIPTION:
The thrust manipulation applies a high velocity and intensity push in a specified direction to correct the position or movement of the sacroiliac joint.

The muscle-energy technique consists of the therapist correcting the sacroiliac joint while the participant is applying active resistance.

For the placebo manipulation, participants will receive a false manipulation over the affected joint, without producing movement at the sacroiliac joint.

ELIGIBILITY:
Inclusion Criteria:

* Amateur runners who perform between 10-30 km per week) and present a sacroiliac joint dysfunction.

Exclusion Criteria:

* Low back pain
* Vertebral bone pathology
* Radicular neurological condition
* Fracture or recent surgical intervention in the lumbosacral or pelvic region
* Anatomical short leg with a difference greater than 0.5 cm
* Pregnant
* Fear of manipulation technique

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Weight Distribution | throughout study completion, an average of 1 month
  The baropodometry platform will be used to measure the distribution of weight (%) between legs.
Center of Gravity Displacement | throughout study completion, an average of 1 month
  The baropodometry platform will measure the distance traveled (mm in x- and y-axis)
Center of Pressure Displacement | throughout study completion, an average of 1 month
  The baropodometry platform will measure the distance traveled (mm in x- and y-axis)
Change in Plantar support | throughout study completion, an average of 1 month
  The baropodometry platform will measure the distribution of weight (%) across the foot (i.e., forefoot and rearfoot)
Foot Plantar Pressure | throughout study completion, an average of 1 month
  The baropodometry platform will measure the points of pressure across the foot with the aid of colorimetry (N/cm2)

CONTACTS AND LOCATIONS:
Overall Officials: Linda H Chung, PhD, Principal Investigator — UCAM Research Center for High Performance Sport
Locations (1):
- UCAM Research Center for High Performance Sport, Guadalupe, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No